CLINICAL TRIAL: NCT07325175
Title: Quantifying Motor Network Dynamics to Predict and Enhance Outcomes in Pediatric Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Travis Larsh, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-9025
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-05

CONDITIONS: Dystonia; Pediatric; Deep Brain Stimulation; Motor Development
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DBS (Experimental): Patients with DBS will complete neurophysiological recordings with DBS on and off
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Subjects with DBS will complete protocol with and without active stimulation

SUMMARY:
The goal of this study is to understand the development and progression of childhood dystonia, a movement disorder, in children. The main questions it aims to answer are:

How does the activity of the neural network evolve in children with dystonia in the context of motor development? What are the effects of chronic and active stimulation on cortical and subcortical motor network function in children with deep brain stimulation (DBS)?

Participants will:

* Undergo noninvasive electrophysiological measurements (EEG, EMG) to quantify neural network activity. They will be tested at rest and during a simple motor reaction task.
* Children with DBS will be assessed in the on and off DBS state to assess effects of chronic and active changes in motor network function.

ELIGIBILITY:
Inclusion Criteria:

* For dystonia subjects:
* Dx of dystonia (with and without DBS)
* willingness and ability to complete study protocols.
* For Typically Developing Controls:
* normal developmental milestones
* absence of any neuropsychiatric disorder
* no significant medical condition.

Exclusion Criteria:

* history of epilepsy
* presence of implanted medical devices (except DBS in dystonia subjects)
* lack of cognitive or physical ability to complete study protocol.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change in Motor Network Aperiodic Activity | -Baseline -Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Longitudinal change in Motor Network Periodic Activity | -Baseline -Through study completion, an average of 2 years
Longitudinal change in Motor Network EEG connectivity | -Baseline -Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon reasonable request and discussion